CLINICAL TRIAL: NCT03774381
Title: Effect of Bifidobacterium Breve B-3 on Body Fat in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-2018-016
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium breve B-3 group (Experimental): 160 mg mg of Bifidobacterium breve B-3 was orally administered per day for 12 weeks.
  Interventions: Dietary Supplement: Bifidobacterium breve B-3
- Control group (Placebo Comparator): 160 mg of placebo was orally administered per day for 12 weeks.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Bifidobacterium breve B-3 — 160 mg of Bifidobacterium breve B-3 is orally administered per day for 12 weeks.
  Arms: Bifidobacterium breve B-3 group
Dietary Supplement: Control group — 160 mg of placebo is orally administered per day for 12 weeks.
  Arms: Control group

SUMMARY:
Comparison of a randomized, double-blind, and control-group study for the effect of oral ingestion of Bifidobacterium breve B-3 on body fat reduction in obese adults

DETAILED DESCRIPTION:
Our aim is to investigate the effect of oral ingestion of Bifidobacterium breve B-3 on body fat reduction in adults by a randomized, double-blind, and control-group study.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27~30 kg/m2

Exclusion Criteria:

* Within the last 6 months, severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.), heart disease(Angina pectoris, myocardial infarction, heart failure, arrhythmia requiring treatment), or malignant diseases (however, although subjects have a history of cerebrovascular disease and heart disease, they can be included if their status are clinically stable)
* Patients with uncontrolled hypertension (blood pressure greater than 160/100 mmHg)
* Diabetic patients with poor glycemic control with a fasting blood glucose of 160 mg/dl or more
* Those who are treated with hypothyroidism or hyperthyroidism
* Creatinine levels: more than twice the normal upper limit
* Aspartate transaminase (AST), Alanine transaminase (ALT) levels: more than twice the normal upper limit
* Those complaining of severe gastrointestinal symptoms such as heartburn and indigestion
* Drugs that affect weight within the last month (absorption inhibitors and Appetite suppressant, health food / supplements related to obesity improvement, psychiatric Drugs, beta blockers, diuretics, birth control pills, steroids, female hormones) If you are taking
* Participated in the commercial obesity program within the last 3 months.
* If you have participated or are planning to participate in another clinical trial within the past month If yes
* Alcohol abuser
* Smoking abstinence within 3 months
* If they are pregnant or lactating or have a pregnancy plan during the clinical trial
* Those with allergic reactions to the constituent food
* Any person deemed inappropriate by the researcher for other reasons

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Body fat | Change from baseline body fat at 12 weeks
  dual energy x-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Integrated Research Institute for Natural Ingredients and Functional Foods, Yangsan, South Korea